CLINICAL TRIAL: NCT04472247
Title: Sedation Monitoring Using Frontal Electroencephalogram, Electromyogram and Hemodynamic Responses to Pain in Critical Care
Status: Completed | Type: Observational
Sponsor: University of Helsinki (Other)
Responsible Party: Principal Investigator, Juhani Akseli Stewart, Dr. Juhani Stewart, MD, University of Helsinki
Other Study IDs: Responsiveness
Record Dates: First submitted 2020-07-11; First posted 2020-07-15 (Actual); Last update posted 2020-07-15 (Actual); Status verified 2020-07

CONDITIONS: Electroencephalography; Critical Care; Electromyography

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Critical Care Patients: Critical care patients requiring mechanical ventilation via an endotracheal tube, with invasive hemodynamic monitoring via an arterial line, and receiving intravenous sedation by continuous infusion (propofol, midazolam).
  Interventions: Diagnostic Test: Continuous EEG and EMG monitoring, with derived variables

INTERVENTIONS:
Diagnostic Test: Continuous EEG and EMG monitoring, with derived variables — All patients are monitored during their ICU stay by frontal EEG and EMG measuring devides, which are already in clinical use.

SUMMARY:
Purpose: Assessing nociception and sedation in mechanically ventilated patients in the ICU is challenging, with few reliable methods available for continuous monitoring. Measurable cardiovascular and neurophysiological variables, such as blood pressure, heart rate, frontal EEG, and frontal EMG, might provide a medium for sedation and nociception monitoring. The hypothesis of this explorative study is that the aforementioned variables correlate with the level of sedation, as described by the Richmond Agitation-Sedation score (RASS).

Methods: Thirty adult postoperative ICU patients on mechanical ventilation and receiving intravenous sedation, excluding patients with primary neurological disorders, head injury, or need for continuous neuromuscular blockage. Continuous measurements of bispectral index (BIS), EMG power (EMG), EMG-derived Responsiveness Index (RI), averaged blood pressure variability (ARV), and Surgical Pleth Index (SPI) were tested against repeated RASS measurements, and separately against responsiveness to painful stimuli at varying RASS levels.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (over 18 years old)
* Postoperative ICU admission (planned and un-planned admissions), on mechanical ventilation via an endotracheal tube, with invasive hemodynamic monitoring via an arterial line
* receiving intravenous sedation by continuous infusion (propofol, midazolam).

Exclusion Criteria:

primary neurological disorders (including stroke, cardiac arrest with probable hypoxic brain injury, intracranial hemorrhage, and head injury with reduced level of consciousness prior to intubation), the continuous use of neuromuscular blocking agents during monitoring, confirmed meningitis or encephalitis, or a short data collection time (less than 12 hours).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Postoperative patients, requiring postoperative critical care.
Sampling Method: Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2007-05-07 (Actual); Primary Completion 2009-04-01 (Actual); Study Completion 2009-04-01 (Actual)

PRIMARY OUTCOMES:
EEG and EMG variables correlate with the level of sedation (as measured by the established RASS score), and are reactive with nociceptive stimulation. | 2 (1-3) days from admission to ICU
  Noninvasive neuromonitoring variables are collected and analysed against the RASS score, which quantifies patient's sedation level.

CONTACTS AND LOCATIONS:
Locations (2):
- Finland (2):
  - Helsinki University Central Hospital, Department of Anesthesiology and Intensive Care, Helsinki, Uudenmaan Lääni
  - Helsinki University Central Hospital, Department of Cardiac Surgery, Helsinki, Uudenmaan Lääni

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Barr J, Fraser GL, Puntillo K, Ely EW, Gelinas C, Dasta JF, Davidson JE, Devlin JW, Kress JP, Joffe AM, Coursin DB, Herr DL, Tung A, Robinson BR, Fontaine DK, Ramsay MA, Riker RR, Sessler CN, Pun B, Skrobik Y, Jaeschke R; American College of Critical Care Medicine. Clinical practice guidelines for the management of pain, agitation, and delirium in adult patients in the intensive care unit. Crit Care Med. 2013 Jan;41(1):263-306. doi: 10.1097/CCM.0b013e3182783b72. PMID 23269131
- [Result] Ball J. How useful is the bispectral index in the management of ICU patients? Minerva Anestesiol. 2002 Apr;68(4):248-51. PMID 12024092
- [Result] Fraser GL, Riker RR. Bispectral index monitoring in the intensive care unit provides more signal than noise. Pharmacotherapy. 2005 May;25(5 Pt 2):19S-27S. doi: 10.1592/phco.2005.25.5_part_2.19s. PMID 15899745